CLINICAL TRIAL: NCT00213239
Title: The Minimum Effective Dose of Remifentanil When Co-administered With Propofol for Lumbar Puncture in Children: A Dose-finding Study
Brief Title: A Dose Finding Study of Remifentanil and Propofol for Lumbar Punctures in Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jason Hayes, Staff Anesthesiologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000007479
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2018-08-10 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Hematologic Diseases; Neoplasms
Keywords: spinal puncture; remifentanil; propofol; anesthesia; dose finding; pediatrics
MeSH Terms: conditions — Hematologic Diseases; Neoplasms | interventions — Remifentanil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol 4 mg/kg group (Experimental): First patient in this arm will receive a bolus of propofol 4 mg/kg followed by remifentanil 0.5 mcg/kg. Subsequent patients randomized to this arm will receive propofol 4 mg/kg but the dose of remifentanil will be determined using the Dixon up-and-down method (i.e. based on the response of the previous patient)
  Interventions: Drug: Remifentanil
- Propofol 2 mg/kg group (Experimental): First patient in this arm will receive a bolus of propofol 2 mg/kg followed by remifentanil 1 mcg/kg. Subsequent patients randomized to this arm will receive propofol 2 mg/kg but the dose of remifentanil will be determined using the Dixon up-and-down method (i.e. based on the response of the previous patient)
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — The first patient in this group will receive 4 mg/kg propofol and 0.5 ug/kg respectively. The dose of remifentanil in subsequent patients will be determined by the Dixon up-and-down method.
  Arms: Propofol 4 mg/kg group
Drug: Remifentanil — The first patient in this group will receive 2 mg/kg propofol and 1.0 ug/kg respectively. The dose of remifentanil in subsequent patients will be determined by the Dixon up-and-down method.
  Arms: Propofol 2 mg/kg group

SUMMARY:
This study will examine whether the combination of two anaesthetic medications, propofol and remifentanil, is suitable for short duration surgical procedures, providing a shorter recovery time and fewer side effects than either drug used alone.

DETAILED DESCRIPTION:
Propofol is the primary medication used by anesthesiologists at HSC to provide sedation for lumbar puncture. Propofol provides amnesia, anxiolysis, and hypnosis, but because propofol has no analgestic properties patients often respond to the pain of LP needle insertion. To ensure patient immobility, the dose of propofol is often increased, resulting in a duration of action that is excessive for lumbar puncture. Remifentanil is an ultra-short acting opioid which can be used to provide analgesia and sedation for short painful procedures with minimal residual pain. However, when used as the sole agent, remifentanil is associated with a high incidence of respiratory depression and/or arterial oxygen desaturation and does not provide amnesia or anxiolysis. The combination of propofol and remifentanil may be particularly suitable for short duration procedures, providing a shorter recovery time and fewer side effects than either drug used alone.

The objective is to determine the minimum effective dose of remifentanil required to prevent movement for insertion of a lumbar puncture needle when co-administered with propofol. The results obtained from this study will be used in a future study of the recovery characteristics of propofol and remifentanil in children undergoing lumbar puncture.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of a hemato-oncological disorder
* Scheduled to undergo a lumbar puncture
* Aged 4-11 years
* Male or female
* Unpremedicated
* Willing and able to provide informed consent (or informed consent by parents)

Exclusion Criteria:

* Children who are known or suspected to be difficult to ventilate by face mask
* Children who are deemed medically unfit to receive either of the two study medications
* Children who are obese (weight for height > 95th percentile,
* Children who do not have an indwelling intravenous line

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2005-09; Primary Completion 2007-09 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hayes, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Result] Hayes JA, Lopez AV, Pehora CM, Robertson JM, Abla O, Crawford MW. Coadministration of propofol and remifentanil for lumbar puncture in children: dose-response and an evaluation of two dose combinations. Anesthesiology. 2008 Oct;109(4):613-8. doi: 10.1097/ALN.0b013e31818629f3. PMID 18813039
- See also: Published October 2008 — http://anesthesiology.pubs.asahq.org/article.aspx?articleid=1922581&resultClick=3

RESULTS

PARTICIPANT FLOW:
Groups:
- Propofol 4 mg/kg: Remifentanil: The first patient in this group will receive 4 mg/kg propofol and 0.5 ug/kg respectively. The dose of remifentanil in subsequent patients will be determined by the Dixon up-and-down method.
- Propofol 2mg/kg: Remifentanil: The first patient in this group will receive 2 mg/kg propofol and 1.0 ug/kg respectively. The dose of remifentanil in subsequent patients will be determined by the Dixon up-and-down method.
Period: Overall Study
Arm/Group | Propofol 4 mg/kg | Propofol 2mg/kg
Started | 32 | 32
Completed | 32 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Propofol 4mg/kg: Remifentanil: The first patient in this group will receive 4 mg/kg propofol and 0.5 ug/kg respectively. The dose of remifentanil in subsequent patients will be determined by the Dixon up-and-down method.
- Total: Total of all reporting groups
Arm/Group | Propofol 4mg/kg | Propofol 2mg/kg | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.6 (2.6) | 5.2 (2.1) | 5.3 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 22 | 19 | 41

OUTCOME MEASURES:

1. Primary Outcome: Dose of Remifentanil Required to Prevent Movement in Response to Lumbar Puncture Needle Insertion
Description: Minimum effective dose (Dixon methodology) and ED98 required to prevent movement during lumbar puncture needle insertion
Time Frame: Movement measured at the time of lumbar puncture needle insertion.
Population: Minimum effective dose of remifentanil to prevent movement during lumbar puncture insertion
Measure: Mean (Standard Deviation); unit: micrograms/kg
Groups:
- 2.0 mg/kg Propofol: Remifentanil: The first patient in this group will receive 2 mg/kg propofol and 1.0 ug/kg respectively. The dose of remifentanil in subsequent patients will be determined by the Dixon up-and-down method.
- 4.0 mg/kg Propofol: Remifentanil: The first patient in this group will receive 4 mg/kg propofol and 0.5 ug/kg respectively. The dose of remifentanil in subsequent patients will be determined by the Dixon up-and-down method.
Arm/Group | 2.0 mg/kg Propofol | 4.0 mg/kg Propofol
Number analyzed (Participants) | 32 | 32
micrograms/kg
  Minimum effective dose | 0.96 (0.23) | 0.28 (0.22)
  ED98 | 1.50 (1.0) | 0.52 (1.06)

2. Secondary Outcome: Incidence of Adverse Events.
Time Frame: Followed for the length of the procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | 2.0 mg/kg Propofol | 4.0 mg/kg Propofol
Number analyzed (Participants) | 32 | 32
Participants
  Bradycardia | 0 | 0
  Hypotension | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from administration of study drugs until discharge from recovery room.
Arm/Group | Propofol 4 mg/kg | Propofol 2mg/kg
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propofol 4 mg/kg (N=32) | Propofol 2mg/kg (N=32)
Bradycardia (General disorders) | 0 (0) | 0 (0)
Hypotension (General disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No